CLINICAL TRIAL: NCT05724433
Title: VIrtual Care To Improve Outcomes and RecoverY From Heart Failure Hospitalization (VICTORY-HF) RCT
Brief Title: VIrtual Care To Improve Outcomes and RecoverY From Heart Failure Hospitalization
Acronym: VICTORY-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Harriette Van Spall, Assistant Professor of Medicine, Division of Cardiology, McMaster University, Population Health Research Institute, Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: VICTORY-HF RCT
Record Dates: First submitted 2019-08-31; First posted 2023-02-13 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Heart Failure
Keywords: Heart Failure; Randomized Controlled Trial; Digital Health; Knowledge Translation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: This is an unblinded parallel multi-center Randomized Controlled Trial (RCT) of virtual HF clinics + routine care versus routine care alone in patients discharged after a hospitalization or urgent/emergency visit for HF. Randomization will be at the level of the patients and stratified by hospital site.
  Patients and clinicians will be unblinded, but those analyzing data will be blinded. We will adopt a pragmatic approach to this study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual HF care (Experimental): Patients will receive virtual HF care to optimize medical therapies
  Interventions: Other: Virtual HF Care
- Routine HF care (Other): Participants will receive routine HF care
  Interventions: Other: Routine HF Care

INTERVENTIONS:
Other: Virtual HF Care — Patients will receive virtual visits for 3 months following hospitalization / emergency department (ED) visit for HF. Physiologic measures will be monitored remotely and therapies will be optimized.
  Arms: Virtual HF care
Other: Routine HF Care — Care as determined by the treating physician
  Arms: Routine HF care

SUMMARY:
The clinic visits (intervention) will continue for 90 days, which represents the follow-up period for the primary medication and health status outcomes. The co-primary clinical outcomes will be obtained at 180 days.

DETAILED DESCRIPTION:
Heart failure (HF) is a leading cause of death, hospitalization, and healthcare system expenditure in Canada. While care in HF clinics - multidisciplinary clinics that focus on optimal management of HF - improves health outcomes in HF, there are disparities in access to such care across our province. To respond to the needs of patients and the health care system, the investigators propose to develop and implement a virtual model of care that will enable Canadians with HF to receive outpatient HF care and medical optimization remotely. The investigators hypothesize that relative to routine care alone, virtual HF clinics will improve a composite of implementation and clinical outcomes.

A pilot phase was conducted to assess the acceptability and feasibility of the intervention, assess change in health status, refine the virtual delivery process and healthcare processes, and use these to finalize protocols and guide the larger clinical trial. Data collection during the pilot phase focused on the process outcomes approved by HiREB (ID 5441).

ELIGIBILITY:
Inclusion Criteria:

Adult patients ≥ 18 years old who:

1. Are being discharged after hospitalization or urgent visit for HF as

   1. a primary diagnosis or
   2. significant complication (prolonging length of stay) of another diagnosis OR Have been referred for an initial consult at a cardiology clinic within 1 week of hospitalization or urgent visit for HF as a primary or secondary diagnosis, as described above.
2. Have left ventricular ejection fraction (LVEF) < 50% within the preceding 3 months.
3. Have NT-proBNP of > 900 pg/ml during hospital admission or within 7 days after discharge from the ED
4. Have a mailing address for patient or caregiver
5. Provide verbal consent

Exclusion Criteria:

1. Died or left hospital before medically advised hospital discharge
2. Unable to self-assess or communicate symptoms (e.g. clinically evident dementia)
3. Unable to engage with digital health technology or follow up
4. Severe valve disease
5. Recipient of or on waiting list for LVAD or cardiac transplant
6. Complex congenital heart disease, hypertrophic obstructive cardiomyopathy, or amyloid cardiomyopathy
7. Severe lung disease with symptoms on minimal exertion, forced expiratory volume during 1 second (FEV1) < 1 litre, severe pulmonary hypertension with RVSP > 60 mm Hg, or on home oxygen
8. Severe kidney disease (persistent eGFR < 30 mL/min/1.73m2)
9. Active malignancy
10. Receiving palliative care or expected life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 891 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary "Hierarchical" Composite Outcome of: | 30 and 90 days
  1. Target dose of BB, ARNI or ACEi/ARB, MRA, and SGLT2i at 90 days
  2. GDMT intensification at 30 days, defined as (a) initiation or up-titration of beta-blocker; (b) switch from another beta blocker to carvedilol, bisoprolol, or extended-release metoprolol; (c) initiation or up-titration of ACEi/ARB or ARNI; (d) switch from ACEi/ARB to ARNI; (e) initiation or up-titration of MRA; or (f) initiation of SGLT2i
  3. Change in health status, as measured by the KCCQ-12 summary score at 90 days
  PLEASE NOTE: THESE ARE "HIERACHIAL OUTCOMES"
Co-primary "Hierarchical" Composite Outcome of: | 90 and 180 days
  1. All cause death at 180 days
  2. HF hospitalization at 180 days
  3. All-cause ED visit at 180 days
  4. Change in KCCQ-12 summary score at 90 days
  PLEASE NOTE: THESE ARE "HIERACHIAL OUTCOMES"

SECONDARY OUTCOMES:
GDMT use | 90 days
  Achievement of at least 50% of the target doses of BB, ACEi/ARB or ARNI, MRA, SGLT2i at 90 days.
Clinical Outcomes | 90 days and 180 days
  i) Time to composite all-cause death, HF hospitalization, or all-cause ED visit at 180 days ii) Components of composite endpoint
  * Time to all-cause death
  * Time to HF hospitalization
  * Time to all-cause ED visit iii) Change in health status (KCCQ-12 summary score) at 90 days
Healthcare utilization | 90 days and 180 days
  i) direct healthcare cost at 90 and 180 days
Healthcare utilization | 90 days and 180 days
  ii) number of virtual and in-person clinic visits per patient in 90 days.

CONTACTS AND LOCATIONS:
Overall Officials: Harriette Van Spall, MD, Principal Investigator — McMaster University
Locations (9):
- Canada (5):
  - St. Joseph's Healthcare Hamilton, Hamilton, Onatrio
  - Hamilton General Hospital, Hamilton, Ontario
  - Juravinski Hospital Cancer Centre, Hamilton, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - Unity Health Toronto, Toronto, Ontario
- Tunisia (4):
  - Fattouma Bourguiba Hospital, Monastir
  - Hedi Chaker Hospital, Sfax
  - Sahloul Hospital, Sousse
  - Military Hospital, Tunis

IPD SHARING:
Plan to Share IPD: No